CLINICAL TRIAL: NCT04949308
Title: High or Low. Nasal Nitric Oxide Across Mutations in Primary Ciliary Dyskinesia. A Genotype/Phenotype Analysis of Nasal NO in Patients With PCD Within the European Reference Network (ERN)
Brief Title: Nasal Nitric Oxide Across Mutations in Primary Ciliary Dyskinesia
Acronym: nNO_PCD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Collaborators: Rigshospitalet, Denmark (Other); Hospital Vall d'Hebron (Other); KU Leuven (Other); Amsterdam UMC, location VUmc (Other); University of Valencia (Other); NOVA Medical School (Other); University of Geneva, Switzerland (Other); University of Bern (Other); Ruhr University of Bochum (Other); Charite University, Berlin, Germany (Other); Hannover Medical School (Other); Medical University of Vienna (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); University College, London (Other); University of Dundee (Other); University of Southampton (Other); University of Leicester (Other); University of Pisa (Other); Federico II University (Other); Bambino Gesù Hospital and Research Institute (Other); University of Nicosia (Other); Oslo University Hospital (Other); Hospital de Niños R. Gutierrez de Buenos Aires (Other); Hacettepe University (Other); Marmara University (Other); University Hospital, Motol (Other); University Children's Hospital, Zurich (Other); The Leeds Teaching Hospitals NHS Trust (Other); Hadassah Medical Organization (Other); Göteborg University (Other); Schneider Children's Medical Center, Israel (Other); University of Sao Paulo (Other); University Hospital of Cologne (Other); University of Belgrade (Other); University Hospital, Martin (Other); Abderrahmane Mami Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: JR_nNO_PCD_09_2020
Record Dates: First submitted 2021-06-24; First posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Ciliary Motility Disorders; Primary Ciliary Dyskinesia
MeSH Terms: conditions — Ciliary Motility Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Genetic diagnosis: Genetic: Genetic diagnosis No Intervention foreseen, but genetically confirmed diagnosis of PCD (bi-allelic mutations in a gene, known to cause PCD) with typical clinical symptoms of PCD and at least one other method confirming PCD-diagnosis is needed

SUMMARY:
Primary Ciliary Dyskinesia (PCD) is a rare genetic disorder characterized by dysfunction of motile cilia associated with recurrent infections of the airways, laterality defects (Situs inversus totalis in about 50% of cases) and fertility problems. At present, mutations in > 45 genes associated with PCD and mucociliary clearance disorders have been identified, representing most likely two thirds of all human cases.

The aims of this study are:

1. Correlation between nasal NO levels and distinct PCD genotypes
2. Determination of further parameters potentially associated with nasal NO levels in genotyped PCD individuals

   1. course of clinical manifestations (e.g. neonatal distress, infections, bronchiectasis)
   2. diagnostic results (HVMA, TEM, IF)
   3. lung function outcome (FVC, FEV1)

DETAILED DESCRIPTION:
Nasal Nitric Oxide (nNO) concentration is usually low or very low in patients with Primary Ciliary Dyskinesia (PCD) for yet unknown reasons (1).

Measured nNO holds a strong ability to separate healthy subjects from patients with PCD in both childhood and adulthood and across several different nNO sampling modalities (2) (3-5) and nNO is widely used as an important supplementary diagnostic test for PCD work up in both Europe (6) and North America (7). Low nNO in PCD was first reported 26 years ago (8). Nasal NO has been associated with host paranasal sinus defense as sufficient nNO production in non-PCD subjects is thought to play a role in maintaining paranasal sinus sterility (9). Furhermore, ciliary beating seems to be upregulated by a NO dependent pathway in bovine airway epithelium (10), influencing mucociliary clearance. However, human in vitro studies of ciliated airway cells in air-liquid-interface (ALI) culture have been ambiguous as to whether the biosynthesis of NO in PCD is impaired (11) (12) or not (13; 14) and the etiology of low nNO in PCD and presumed link to ciliary beating remains unclear. So far, attempts to link PCD phenotype and genotype has indicated that patients with PCD harboring CCDC39 and CCDC40 mutations may have a poorer lung function development (15).

In rare cases of PCD (<5%) (16) nNO concentration is within normal range. More than 14 different PCD-causing genes (e.g RSPH1, GAS8, RPGR, CCNO, CCDC103, CFAP221, DNAH9, FOXJ1, GAS2L2, LRRC56, NEK10, SPEF2, STK36, TTC12) has been associated with nNO values above the agreed cut off for nNO-production rate of 77 nL/min in a few patients with PCD (16). However, individuals with NEK10 or FOXJ1 mutations, for example, display a very severe respiratory phenotype (17), but making a diagnosis is challenging because of normal nNO values as well as apparently normal ciliary beating.

Since nNO also holds potential as an outcome parameter in future clinical trials of PCD, better understanding of nNO in PCD is warranted.

Demand of large number of patients with PCD is crucial, keeping the rareness of nearnormal and normal nNO levels in PCD in mind. Motivated by the analysis of lung function in a large cohort of genotyped PCD-patients, this multicenter Involvement across international PCD centers is an obvious opportunity for gaining such further knowledge with the focus on nasal NO.

The aims of this study are:

1. Correlation between nasal NO levels and distinct PCD genotypes
2. Determination of further parameters potentially associated with nasal NO levels in genotyped PCD individuals

   1. course of clinical manifestations (e.g. neonatal distress, infections, bronchiectasis)
   2. diagnostic results (HVMA, TEM, IF)
   3. lung function outcome (FVC, FEV1)

Inclusion criteria:

1. Patients with a genetically confirmed diagnosis of PCD (bi-allelic mutations in a gene, known to cause PCD) with typical clinical symptoms of PCD
2. PCD individuals of all age groups with at least one nNO measurement performed according to diagnostic guidelines. Serial nNO measurements should be included if available (e.g. yearly), at least for infants and young children

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a genetically confirmed diagnosis of PCD (bi-allelic mutations in a gene, known to cause PCD) with typical clinical symptoms of PCD
2. PCD individuals of all age groups with at least one nNO measurement performed according to diagnostic guidelines. Serial nNO measurements should be included if available (e.g. yearly), at least for infants and young children

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a genetically confirmed diagnosis of PCD (bi-allelic mutations in a gene, known to cause PCD) with typical clinical symptoms of PCD
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Genotype-nasal Nitric Oxide Corelation | up to 20 years retrospective
  nNO in correlation to the genetic make-up

CONTACTS AND LOCATIONS:
Overall Officials: Heymut Omran, Prof,Dr,MD, Study Chair — University Hospital Muenster
Locations (1):
- University Hospital Münster, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided